CLINICAL TRIAL: NCT03477461
Title: Effects of Terlipressin on Management of Potential Organ Donors：a Retrospective Study
Brief Title: Effects of Terlipressin on Management of Potential Organ Donors
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Effects of terlipressin
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Organ Donors
MeSH Terms: interventions — Terlipressin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- terlipressin group: patients presented with oliguria or high levels creatinine
  Interventions: Drug: terlipressin

INTERVENTIONS:
Drug: terlipressin — a continuous infusion of terlipressin (0.4 mg/kg/h) was initiated

SUMMARY:
During brain death, many significant systemic changes take place and among these, the most notable is hemodynamic instability.

In the pathogenesis of brain death, after the hypertensive phase of the "catecholamine storm", arterial tonus and heart inotropism eventually deteriorate, leading to hypotension and hypoperfusion. Therefore, vasopressor agents are necessary in treatment of brain-dead organ donors. The most commonly used and recommended vasoactive drugs for this indication are dopamine, norepinephrine, and vasopressin.The Transplantation Committee of the American College of Cardiology recommends vasopressin as the primary vasoactive drug for treating hemodynamic instability and diabetes insipidus in brain-death heart donors.

Terlipressin (TP) is a new type of synthetic long-acting vasopressin preparations, AVP long-acting derivatives, belongs to a kind of precursor drugs, itself is inactive, the body through the aminopeptidase, slow "release" of a reactive lysine vasopressin. On the one hand，terlipressin can splanchnic vascular smooth muscle contraction, reduces splanchnic blood flow (e.g., reduce blood flow to the mesenteric, spleen, uterus, etc), to ensure the flow of blood to the important viscera;On the other hand, it reduces the concentration of plasma renin, increases the perfusion of renal blood flow, and improves the glomerular filtration rate, thus improving renal function.From the pharmacological perspective, it is better than arginine vasopressin for the stability of hemodynamics and the perfusion of tissue.

Whether or not it has therapeutic effect on the potential brain death donor with unstable hemodynamics is not studied in the literature at home and abroad.This paper discusses the application value of terlipressin in the management of potential brain death, and provides clinical evidence for the maintenance of brain death donor.

DETAILED DESCRIPTION:
Thermodilution cardiac output was measured in triplicate. Hemodynamic parameters were calculated according to standard formulas.Oxygen delivery index (IDO2) was calculated as arterial oxygen content multiplied by CI. Systemic vascular resistance index (SVRI) was calculated as the MAP minus right atrial pressure divided by CI and multiplied by 80. Pulmonary vascular resistance index (PVRI) was calculated as the mean pulmonary artery pressure (PAP) minus pulmonary artery occlusion pressure divided by CI. Left and right ventricular stroke work index (L and RVSWI) were calculated .The following laboratory parameters were collected: bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT),prothrombin time, and thrombocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-60 years old, gender is not limited, accord with brain death standard patient.
2. Complete ethical procedures, have entered the donation procedure and successful donation.

3 oliguria or high creatinine.

Exclusion Criteria:

1. Patients with uremia.
2. Patients with diabetes.
3. There is known to be an allergy to trelin.
4. Previous patients with coronary heart disease.
5. Active digestive tract hemorrhage, liver dysfunction (Child C), severe 6.coagulation dysfunction, and cannot be corrected, or other specific contraindication.

7.Active HIV infection or HIV, mental disorder, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18 patients were enrolled. All were potential organ donors.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
creatinine | Change from Baseline, 24 hours, 72 hours to Before organ procurement
  Laboratory values

SECONDARY OUTCOMES:
urine volume | Change from Baseline, 24 hours, 72 hours to Before organ procurement
  observed data
glomerular filtration rate | Change from Baseline, 24 hours, 72 hours to Before organ procurement
  Laboratory values
endogenous creatinine clearance rate | Change from Baseline, 24 hours, 72 hours to Before organ procurement
  Laboratory values
Norepinephrine dose | Change from Baseline, 24 hours, 72 hours to Before organ procurement
  monitoring data

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Tai, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No